CLINICAL TRIAL: NCT01029912
Title: Contralaterally Controlled NMES in Chronic Ankle Dorsiflexor Paresis After Stroke
Brief Title: Electrical Stimulation for Recovery of Ankle Dorsiflexion in Chronic Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jayme Knutson, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD061593 (NIH); R21HD061593 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Stroke; Hemiparesis; Lower Extremity Paresis
Keywords: Stroke; Hemiplegia; Footdrop; Electrical Stimulation; Motor Relearning; Neuroplasticity
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- CCNMES (Experimental): Contralaterally Controlled Neuromuscular Electrical Stimulation (CCNMES) Electrical Stimulator
  Interventions: Device: Electrical stimulator
- Cyclic NMES (Active Comparator): Cyclic Neuromuscular Electrical Stimulation (NMES) Electrical Stimulator
  Interventions: Device: Electrical stimulator

INTERVENTIONS:
Device: Electrical stimulator — 6-week intervention
  15 minutes of therapist-guided stimulated ankle exercise + 30 minutes of physical therapy in the laboratory twice a week.
  Self-administered active repetitive ankle dorsiflexion exercise performed twice a day, 6 days a week at home using the device.

SUMMARY:
Ankle dorsiflexor weakness (paresis) is one of the most frequently persisting consequences of stroke. The purpose of this exploratory study is to compare two different treatments -- Contralaterally Controlled Neuromuscular Electrical Stimulation (CCNMES) and Cyclic Neuromuscular Electrical Stimulation (cNMES) -- for improved recovery of ankle movement and better walking after stroke.

DETAILED DESCRIPTION:
Ankle dorsiflexor weakness results in inefficient and unstable gait. While routine physical therapy is beneficial, for many individuals it remains limited in its effectiveness, and consequently many stroke survivors have difficulty walking safely or remain non-ambulatory. Ankle-foot-orthoses (AFOs) are often prescribed to provide ankle stability, but because they limit ankle mobility they may actually inhibit recovery of dorsiflexion. Advanced rehabilitation techniques that emphasize active, repetitive, goal-oriented movement of the impaired limb have produced measurable functional improvements, yet a significant degree of lower extremity disability often remains. In addition, some of these emerging therapies are difficult to administer and are applicable only to patients who retain at least some degree of ambulation. Thus, there is a need for alternative treatments.

This is an exploratory study of an innovative neuromuscular electrical stimulation (NMES) treatment for restoring lower extremity motor control following stroke. We will investigate whether stroke survivors with chronic footdrop recover voluntary ankle dorsiflexion after a novel treatment of NMES. Surface electrodes will deliver stimulation to dorsiflex the ankle with an intensity that is proportional to the amount of dorsiflexion of the other unimpaired ankle. Thus, voluntary dorsiflexion of the unaffected ankle produces stimulated dorsiflexion of the affected ankle. We refer to this stimulation paradigm as Contralaterally Controlled Neuromuscular Electrical Stimulation (CCNMES). In contrast to existing peroneal nerve stimulators, CCNMES is not intended to be used to assist ambulation; rather it is intended as solely a motor retraining paradigm that may reduce lower extremity impairment and improve ambulation. The primary objective of the proposed study is to obtain pilot data so that an estimate can be made of the efficacy of CCNMES in reducing lower extremity impairment and improving ambulation.

Twenty-six chronic stroke survivors (>6 months post-stroke) will be randomized to either CCNMES or cyclic NMES, an intervention that provides electrical stimulation of the ankle dorsiflexors, but with preprogrammed timing and intensity. For both groups, the treatment will last 6 weeks. Assessments of ankle impairment and ambulation will be made at baseline and at end of treatment.

This study is the first randomized controlled trial of CCNMES for restoring ankle dorsiflexion in patients with chronic hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 80 years
* >6 months from a first clinical non-hemorrhagic or hemorrhagic stroke
* Medically stable
* Unilateral lower extremity hemiparesis
* Ankle dorsiflexor strength of ≤4/5 on the Medical Research Council (MRC) scale, while seated
* Able to ambulate 16 feet (5 meters) continuously with minimal assistance or less, without the use of an ankle-foot orthosis (AFO).
* AFO is clinically indicated (footdrop during ambulation or inefficient gait patterns)
* Neuromuscular electrical stimulation (NMES) of the paretic ankle dorsiflexors produces ankle dorsiflexion to neutral without pain.
* Full voluntary dorsiflexion of the contralateral ankle
* Skin intact on hemiparetic lower extremity
* Able to don the NMES system or caregiver available to assist with device if needed.
* Able to hear and respond to stimulator auditory cues
* Able to follow 3-stage commands
* Able to recall 2 of 3 items after 30 minutes

Exclusion Criteria:

* Brainstem stroke
* Severely impaired cognition and communication
* History of peroneal nerve injury
* History of Parkinson's, spinal cord injury, traumatic brain injury, or multiple sclerosis
* Uncontrolled seizure disorder
* Uncompensated hemi-neglect (extinguishing to double simultaneous stimulation)
* Edema of the affected lower extremity
* Absent sensation of lower leg and foot
* Evidence of deep venous thrombosis or thromboembolism
* History of cardiac arrhythmias with hemodynamic instability
* Cardiac pacemaker or other implanted electronic system
* Botulinum toxin injections to any lower extremity muscle in the last 3 months
* Pregnancy
* Currently receiving Physical Therapy for the lower extremity

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayme S. Knutson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nudo RJ, Wise BM, SiFuentes F, Milliken GW. Neural substrates for the effects of rehabilitative training on motor recovery after ischemic infarct. Science. 1996 Jun 21;272(5269):1791-4. doi: 10.1126/science.272.5269.1791. PMID 8650578
- [Background] Luft AR, McCombe-Waller S, Whitall J, Forrester LW, Macko R, Sorkin JD, Schulz JB, Goldberg AP, Hanley DF. Repetitive bilateral arm training and motor cortex activation in chronic stroke: a randomized controlled trial. JAMA. 2004 Oct 20;292(15):1853-61. doi: 10.1001/jama.292.15.1853. PMID 15494583
- [Background] Robbins SM, Houghton PE, Woodbury MG, Brown JL. The therapeutic effect of functional and transcutaneous electric stimulation on improving gait speed in stroke patients: a meta-analysis. Arch Phys Med Rehabil. 2006 Jun;87(6):853-9. doi: 10.1016/j.apmr.2006.02.026. PMID 16731222
- [Background] Rushton DN. Functional electrical stimulation and rehabilitation--an hypothesis. Med Eng Phys. 2003 Jan;25(1):75-8. doi: 10.1016/s1350-4533(02)00040-1. PMID 12485788
- [Background] Khaslavskaia S, Sinkjaer T. Motor cortex excitability following repetitive electrical stimulation of the common peroneal nerve depends on the voluntary drive. Exp Brain Res. 2005 May;162(4):497-502. doi: 10.1007/s00221-004-2153-1. Epub 2005 Feb 9. PMID 15702321
- [Background] Knutson JS, Harley MY, Hisel TZ, Chae J. Improving hand function in stroke survivors: a pilot study of contralaterally controlled functional electric stimulation in chronic hemiplegia. Arch Phys Med Rehabil. 2007 Apr;88(4):513-20. doi: 10.1016/j.apmr.2007.01.003. PMID 17398254
- [Background] Knutson JS, Hisel TZ, Harley MY, Chae J. A novel functional electrical stimulation treatment for recovery of hand function in hemiplegia: 12-week pilot study. Neurorehabil Neural Repair. 2009 Jan;23(1):17-25. doi: 10.1177/1545968308317577. Epub 2008 Sep 23. PMID 18812432
- [Background] Sheffler LR, Hennessey MT, Naples GG, Chae J. Peroneal nerve stimulation versus an ankle foot orthosis for correction of footdrop in stroke: impact on functional ambulation. Neurorehabil Neural Repair. 2006 Sep;20(3):355-60. doi: 10.1177/1545968306287925. PMID 16885421
- See also: Cleveland Functional Electrical Stimulation Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438

RESULTS

PARTICIPANT FLOW:
Groups:
- CCNMES: Contralaterally Controlled Neuromuscular Electrical Stimulation (Electrical Stimulator)
  CCFES Electrical Stimulator: 6-week intervention
  Home: Self-administered active repetitive CCNMES-mediated ankle dorsiflexion exercise performed ten 51-minute sessions (three 15-min sets separated by 3-min rest) per week at home.
  Lab: 15 minutes of therapist-guided CCFES-mediated ankle exercise + 30 minutes of gait training in the laboratory twice a week.
- Cyclic NMES: Cyclic Neuromuscular Electrical Stimulation (Electrical Stimulator)
  Cyclic NMES Electrical Stimulator: 6-week intervention
  Home: Self-administered active repetitive Cyclic NMES-mediated ankle dorsiflexion exercise performed ten 51-minute sessions (three 15-min sets separated by 3-min rest) per week at home.
  Lab: 15 minutes of therapist-guided Cyclic NMES-mediated ankle exercise + 30 minutes of gait training in the laboratory twice a week.
Period: Overall Study
Arm/Group | CCNMES | Cyclic NMES
Started | 14 | 12
Completed | 12 | 12
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Only participants who completed treatment were analyzed.
Groups:
- CCNMES: Contralaterally Controlled Neuromuscular Electrical Stimulation (Electrical Stimulator)
  Electrical stimulator: 6-week intervention
  15 minutes of therapist-guided stimulated ankle exercise + 30 minutes of physical therapy in the laboratory twice a week.
  Self-administered active repetitive ankle dorsiflexion exercise performed twice a day, 6 days a week at home using the device.
- Cyclic NMES: Cyclic Neuromuscular Electrical Stimulation (Electrical Stimulator)
  Electrical stimulator: 6-week intervention
  15 minutes of therapist-guided stimulated ankle exercise + 30 minutes of physical therapy in the laboratory twice a week.
  Self-administered active repetitive ankle dorsiflexion exercise performed twice a day, 6 days a week at home using the device.
- Total: Total of all reporting groups
Arm/Group | CCNMES | Cyclic NMES | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (13.7) | 59.3 (9.1) | 58.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years Since Stroke [Mean (Standard Deviation); unit: years] | 2.7 (1.8) | 3.6 (3.9) | 3.1 (3.0)
Lower Extremity Fugl-Meyer Score [Mean (Standard Deviation); unit: units on a scale] — The Lower Extremity Fugl-Meyer (LEFM) Assessment measures lower limb motor impairment. Participants are asked to attempt to perform isolated and simultaneous movements of the hip, knee, and ankle. Each movement attempt is graded on a 3-point ordinal scale (0, cannot perform; 1, perform partially; and 2, perform fully). These subscores are summed to provide a maximum score of 34, minimum score of 0. Higher scores are considered to be a better outcome.
  units on a scale | 19.1 (6.8) | 18.9 (7.0) | 19.0 (6.8)
Time to complete Modified Emory Functional Ambulation Profile (MEFAP) in seconds [Mean (Standard Deviation); unit: seconds] — The MEFAP is a measure of functional ambulation, measuring the time to ambulate through 5 common environmental terrains: 1) 5-meter walk on a hard floor, 2) 5-meter walk on a carpeted floor, 3) rise from a chair, 3-meter walk, return to seated position, 4) standardized obstacle course (bricks to step over), 5) stair ascent and descent. The five times subscores were added to derive a total time. Lower times are considered to be a better outcome.
  seconds | 120.7 (86.3) | 118.6 (86.5) | 119.7 (84.5)
Gait velocity (cm/sec) [Mean (Standard Deviation); unit: cm/sec] — Gait velocity was assessed using a motion capture and analysis system which collected spatio-temporal data as the participant walked 5-meters 10 times at a self-selected comfortable speed within the field of view of the motion capture system. A higher gait velocity is considered to be a better outcome.
  cm/sec | 39.9 (22.3) | 38.3 (19.1) | 39.1 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Extremity Fugl-Meyer Score at End of Treatment
Description: The Lower Extremity Fugl-Meyer (LEFM) Assessment is a measure of lower limb motor impairment. Participants are asked to attempt to perform a list of isolated and simultaneous movements of the hip, knee, and ankle that take into account synergy patterns, isolated strength, coordination, and hypertonia. Each movement attempt is graded on a 3-point ordinal scale (0, cannot perform; 1, perform partially; and 2, perform fully) and these subscores are summed to provide a maximum score of 34, minimum score of 0.
  Higher scores are considered to be a better outcome. For each individual, the score prior to treatment was subtracted from the score at end of the 6-week treatment. Then for each treatment group, these change scores were averaged.
Time Frame: 2 timepoints: Prior to treatment, and End of treatment at 6 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 12 | 12
units on a scale | 0.93 (0.65) | 1.8 (0.77)

2. Primary Outcome: Change in Gait Velocity (cm/Sec) at End of Treatment
Description: Gait velocity was assessed using a motion capture and analysis system which collected spatio-temporal data as the participant walked 5-meters 10 times at a self-selected comfortable speed within the field of view of the motion capture system. A higher gait velocity is considered to be a better outcome. For each individual, the gait velocity prior to treatment was subtracted from the gait velocity at end of the 6-week treatment. Then for each treatment group, these change values were averaged.
Time Frame: 2 timepoints: Prior to treatment, and End of treatment at 6 weeks.
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 12 | 12
cm/sec | 3.0 (2.1) | 1.2 (2.6)

3. Primary Outcome: Change in Time (Sec) to Complete the Modified Emory Functional Ambulation Profile (MEFAP).
Description: The MEFAP is a measure of functional ambulation, measuring the time to ambulate through 5 common environmental terrains: 1) 5-meter walk on a hard floor, 2) 5-meter walk on a carpeted floor, 3) rise from a chair, 3-meter walk, return to seated position, 4) standardized obstacle course (bricks to step over), 5) stair ascent and descent. The five times subscores were added to derive a total time.
  Lower times are considered to be a better outcome.
  For each individual, the MEFAP completion time prior to treatment was subtracted from the MEFAP completion time at end of the 6-week treatment. Then for each treatment group, these change values were averaged.
Time Frame: 2 timepoints: Prior to treatment, and End of treatment at 6 weeks.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 12 | 12
seconds | -9.6 (2.6) | -3.2 (4.1)

ADVERSE EVENTS:
Arm/Group | CCNMES | Cyclic NMES
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCNMES (N=12) | Cyclic NMES (N=12)
Discomfort from stimulation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No